CLINICAL TRIAL: NCT03377751
Title: Does VoltagE Guided Additional Ablation Improve Procedural Outcome of Atrial Fibrillation Ablation? (The VEGA-AF Study)
Brief Title: Does VoltagE Guided Additional Ablation Improve Procedural Outcome of Atrial Fibrillation Ablation?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Majority of enrolled patients have withdrawn.
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Hong Euy Lim, MD, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUGH17287 (VEGA-AF)
Record Dates: First submitted 2017-12-09; First posted 2017-12-19 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Atrial Fibrillation
Keywords: Catheter ablation; Atrial fibrillation; Low voltage area
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Additional posterior wall isolation (Experimental): Operator will perform pulmonary vein isolation (PVI) and additional posterior wall isolation if low voltage area exists more than 10% of the left atrium
  Interventions: Procedure: Additional posterior wall isolation
- Voltage-guided substrate homogenization (Experimental): Operator will perform pulmonary vein antrum isolation (PVI) and additional substrate modification based on the degree of low voltage area.
  Interventions: Procedure: Voltage-guided substrate homogenization
- PVI only group (Active Comparator): Operator will perform PVI only
  Interventions: Procedure: PVI only group

INTERVENTIONS:
Procedure: Additional posterior wall isolation — PVI and additional posterior wall isolation will be performed according to the following protocol which is based on low voltage area.
  1. Proportion of low voltage area to area of left atrium body <10% : PVI only
  2. Proportion of low voltage area to area of left atrium body ≥10% : PVI + Posterior wall isolation
     * Low voltage area will be measured from more than 1000 points of sampled voltage value during sinus rhythm using PentaRay catheter with 3D mapping system of CARTO (Biosense Webster, CA, USA).
  Arms: Additional posterior wall isolation
Procedure: Voltage-guided substrate homogenization — PVI and additional substrate modification at low voltage areas will be performed according to the following protocol which is based on low voltage area.
  1. Proportion of low voltage area to area of left atrium body <10% : PVI only
  2. Proportion of low voltage area to area of left atrium body ≥10% : PVI + substrate homogenization at low voltage areas
     * Low voltage area will be measured from more than 1000 points of sampled voltage value during sinus rhythm using PentaRay catheter with 3D mapping system of CARTO (Biosense Webster, CA, USA).
  Arms: Voltage-guided substrate homogenization
Procedure: PVI only group — PVI will be performed in this arm.
  Arms: PVI only group

SUMMARY:
This study is designed to investigate whether pulmonary vein isolation(PVI) plus stepwise additional ablation approach based on the degree of low voltage area versus PVI only can improve procedure outcome in persistent atrial fibrillation(AF) patients.

DETAILED DESCRIPTION:
Catheter ablation of AF is well accepted and widely performing treatment method of AF at present. Pulmonary vein isolation (PVI) which aims to electrical isolation of pulmonary veins is currently the standard therapy for AF. But some researchers proposed additional ablation strategy for persistent AF (PeAF) because abnormal atrial substrate may play a role in these patients.

However, there are inconsistent reports regarding a success rate of additional catheter ablation methods other than PVI. Thus, there still is no consensus on which strategy is appropriate in addition to PVI. One of these proposed options is complex fractioned atrial electrograms (CFAE) ablation. A meta-analysis of controlled trials comparing PVI alone versus PVI with CFAE reported that the addition of CFAE ablation results in a statistically significant increase in success rate for PeAF patients. Conversely, a prospective multicenter trial, The Substrate and Trigger Ablation for Reduction of Atrial Fibrillation Trial Part II (STAR-AF II) trial showed that recurrence rate of AF following catheter ablation treatment was not significantly reduced when either linear ablation or ablation of CFAE was performed in addition to PVI. The investigators have previously reported that posterior wall isolation in addition to PVI plus linear lesions reduced recurrence of AF following catheter ablation compared to PVI only but the long-term success rate were markedly lower in the CFAE-guide ablation in addition PVI plus linear lesions group than in PVI plus linear lesions group among PeAF patients. Although benefit of addition CFAE could be originated from modification of abnormal atrial substrate which is generated by structural and electrical remodeling, this possible benefit could be counterbalanced by increased formation of transmural ablation scar which may result in dysfunction of left atrium and recurrence of atrial tachyarrhythmia. A recent study have showed that extent of myocardial injury by catheter ablation was associated with left atrium functional deterioration in patients with paroxysmal AF and myocardial damage provoked that may contribute to recurrence of AF following catheter ablation.

Therefore, identification of PeAF patients who would benefit from additional ablation and tailored stepwise approach based on the identification may lead to reduction of iatrogenic myocardial injury and optimization of the result for the AF catheter ablation.

Recent data have shown that voltage guided mapping of left atrium is a powerful predictor of AF recurrence after PAI and voltage based ablation strategy showed promising result in terms of tailored approach. But, prospective, randomized clinical studies are needed to compare the result of a voltage-based AF ablation to the result of established strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing first-time catheter ablation for AF.
* Willing and able to provide informed consent
* Age greater than or equal to 18 years.

Exclusion Criteria:

* Patients who have previously undergone AF ablation
* Patients with more than mild mitral valve stenosis or mechanical mitral valve replacement
* Patients with chronic renal impairment with creatinine clearance rate of <30 mL/min
* Patients who are pregnant

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Freedom rate of any atrial tachy-arrhythmia during 1 year after ablation procedure | Within 1 year after the ablation procedure
  Any recurrence of ECG or Holter documented atrial tachyarrhythmia*
  * Sustained AF or atrial tachycardia >30 s duration.

SECONDARY OUTCOMES:
Procedure related complication rate | during procedure and follow-up period(up to 1 year)
  any adverse events
Total procedural time | During procedure
  total cumulative amount of radiation exposure

CONTACTS AND LOCATIONS:
Overall Officials: Hong Euy Lim, MD, Ph.D., Principal Investigator — Professor
Locations (3):
- South Korea (3):
  - Korea University Guro Hospital, Seoul, Guro-gu
  - Korea University Anam Hospital, Seoul, Seongbuk-gu
  - Bucheon Sejong Hospital, Bucheon-si

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nattel S, Shiroshita-Takeshita A, Brundel BJ, Rivard L. Mechanisms of atrial fibrillation: lessons from animal models. Prog Cardiovasc Dis. 2005 Jul-Aug;48(1):9-28. doi: 10.1016/j.pcad.2005.06.002. PMID 16194689
- [Background] Reant P, Lafitte S, Jais P, Serri K, Weerasooriya R, Hocini M, Pillois X, Clementy J, Haissaguerre M, Roudaut R. Reverse remodeling of the left cardiac chambers after catheter ablation after 1 year in a series of patients with isolated atrial fibrillation. Circulation. 2005 Nov 8;112(19):2896-903. doi: 10.1161/CIRCULATIONAHA.104.523928. Epub 2005 Oct 31. PMID 16260634
- [Background] Cox JL, Schuessler RB, Lappas DG, Boineau JP. An 8 1/2-year clinical experience with surgery for atrial fibrillation. Ann Surg. 1996 Sep;224(3):267-73; discussion 273-5. doi: 10.1097/00000658-199609000-00003. PMID 8813255
- [Background] Miyazaki S, Kuwahara T, Takahashi A, Kobori A, Takahashi Y, Nozato T, Hikita H, Sato A, Aonuma K, Hirao K, Isobe M. Effect of left atrial ablation on the quality of life in patients with atrial fibrillation. Circ J. 2008 Apr;72(4):582-7. doi: 10.1253/circj.72.582. PMID 18362429
- [Background] Stabile G, Bertaglia E, Senatore G, De Simone A, Zoppo F, Donnici G, Turco P, Pascotto P, Fazzari M, Vitale DF. Catheter ablation treatment in patients with drug-refractory atrial fibrillation: a prospective, multi-centre, randomized, controlled study (Catheter Ablation For The Cure Of Atrial Fibrillation Study). Eur Heart J. 2006 Jan;27(2):216-21. doi: 10.1093/eurheartj/ehi583. Epub 2005 Oct 7. PMID 16214831
- [Background] Haegeli LM, Calkins H. Catheter ablation of atrial fibrillation: an update. Eur Heart J. 2014 Sep 21;35(36):2454-9. doi: 10.1093/eurheartj/ehu291. Epub 2014 Jul 22. PMID 25053659
- [Background] Elayi CS, Verma A, Di Biase L, Ching CK, Patel D, Barrett C, Martin D, Rong B, Fahmy TS, Khaykin Y, Hongo R, Hao S, Pelargonio G, Dello Russo A, Casella M, Santarelli P, Potenza D, Fanelli R, Massaro R, Arruda M, Schweikert RA, Natale A. Ablation for longstanding permanent atrial fibrillation: results from a randomized study comparing three different strategies. Heart Rhythm. 2008 Dec;5(12):1658-64. doi: 10.1016/j.hrthm.2008.09.016. Epub 2008 Sep 17. PMID 19084800
- [Background] Di Biase L, Burkhardt JD, Mohanty P, Sanchez J, Mohanty S, Horton R, Gallinghouse GJ, Bailey SM, Zagrodzky JD, Santangeli P, Hao S, Hongo R, Beheiry S, Themistoclakis S, Bonso A, Rossillo A, Corrado A, Raviele A, Al-Ahmad A, Wang P, Cummings JE, Schweikert RA, Pelargonio G, Dello Russo A, Casella M, Santarelli P, Lewis WR, Natale A. Left atrial appendage: an underrecognized trigger site of atrial fibrillation. Circulation. 2010 Jul 13;122(2):109-18. doi: 10.1161/CIRCULATIONAHA.109.928903. Epub 2010 Jul 6. PMID 20606120
- [Background] Hayward RM, Upadhyay GA, Mela T, Ellinor PT, Barrett CD, Heist EK, Verma A, Choudhry NK, Singh JP. Pulmonary vein isolation with complex fractionated atrial electrogram ablation for paroxysmal and nonparoxysmal atrial fibrillation: A meta-analysis. Heart Rhythm. 2011 Jul;8(7):994-1000. doi: 10.1016/j.hrthm.2011.02.033. Epub 2011 Mar 10. PMID 21397045
- [Background] Verma A, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P; STAR AF II Investigators. Approaches to catheter ablation for persistent atrial fibrillation. N Engl J Med. 2015 May 7;372(19):1812-22. doi: 10.1056/NEJMoa1408288. PMID 25946280
- [Background] Kim JS, Shin SY, Na JO, Choi CU, Kim SH, Kim JW, Kim EJ, Rha SW, Park CG, Seo HS, Oh DJ, Hwang C, Lim HE. Does isolation of the left atrial posterior wall improve clinical outcomes after radiofrequency catheter ablation for persistent atrial fibrillation?: A prospective randomized clinical trial. Int J Cardiol. 2015 Feb 15;181:277-83. doi: 10.1016/j.ijcard.2014.12.035. Epub 2014 Dec 11. PMID 25535691
- [Background] Han SW, Shin SY, Im SI, Na JO, Choi CU, Kim SH, Kim JW, Kim EJ, Rha SW, Park CG, Seo HS, Oh DJ, Hwang C, Lim HE. Does the amount of atrial mass reduction improve clinical outcomes after radiofrequency catheter ablation for long-standing persistent atrial fibrillation? Comparison between linear ablation and defragmentation. Int J Cardiol. 2014 Jan 15;171(1):37-43. doi: 10.1016/j.ijcard.2013.11.041. Epub 2013 Nov 23. PMID 24315152
- [Background] Gibson DN, Di Biase L, Mohanty P, Patel JD, Bai R, Sanchez J, Burkhardt JD, Heywood JT, Johnson AD, Rubenson DS, Horton R, Gallinghouse GJ, Beheiry S, Curtis GP, Cohen DN, Lee MY, Smith MR, Gopinath D, Lewis WR, Natale A. Stiff left atrial syndrome after catheter ablation for atrial fibrillation: clinical characterization, prevalence, and predictors. Heart Rhythm. 2011 Sep;8(9):1364-71. doi: 10.1016/j.hrthm.2011.02.026. Epub 2011 Feb 23. PMID 21354332
- [Background] Wu SH, Jiang WF, Gu J, Zhao L, Wang YL, Liu YG, Zhou L, Gu JN, Xu K, Liu X. Benefits and risks of additional ablation of complex fractionated atrial electrograms for patients with atrial fibrillation: a systematic review and meta-analysis. Int J Cardiol. 2013 Oct 25;169(1):35-43. doi: 10.1016/j.ijcard.2013.08.083. Epub 2013 Sep 7. PMID 24083885
- [Background] Kim JS, Im SI, Shin SY, Kang JH, Na JO, Choi CU, Kim SH, Kim EJ, Rha SW, Park CG, Seo HS, Oh DJ, Hwang C, Kim YH, Yong HS, Lim HE. Changes in Left Atrial Transport Function in Patients Who Maintained Sinus Rhythm After Successful Radiofrequency Catheter Ablation for Atrial Fibrillation: A 1-Year Follow-Up Multislice Computed Tomography Study. J Cardiovasc Electrophysiol. 2017 Feb;28(2):167-176. doi: 10.1111/jce.13128. Epub 2016 Dec 15. PMID 27859888
- [Background] Lim HE, Choi CU, Na JO, Choi JI, Kim SH, Kim JW, Kim EJ, Han SW, Park SW, Rha SW, Park CG, Seo HS, Oh DJ, Hwang C, Kim YH. Effects of iatrogenic myocardial injury on coronary microvascular function in patients undergoing radiofrequency catheter ablation of atrial fibrillation. Circ Arrhythm Electrophysiol. 2013 Apr;6(2):318-26. doi: 10.1161/CIRCEP.113.000282. Epub 2013 Mar 9. PMID 23476035
- [Background] Rolf S, Kircher S, Arya A, Eitel C, Sommer P, Richter S, Gaspar T, Bollmann A, Altmann D, Piedra C, Hindricks G, Piorkowski C. Tailored atrial substrate modification based on low-voltage areas in catheter ablation of atrial fibrillation. Circ Arrhythm Electrophysiol. 2014 Oct;7(5):825-33. doi: 10.1161/CIRCEP.113.001251. Epub 2014 Aug 23. PMID 25151631
- [Background] Rolf S, Hindricks G, Sommer P, Richter S, Arya A, Bollmann A, Kosiuk J, Koutalas E. Electroanatomical mapping of atrial fibrillation: Review of the current techniques and advances. J Atr Fibrillation. 2014 Dec 31;7(4):1140. doi: 10.4022/jafib.1140. eCollection 2014 Dec. PMID 27957132
- [Background] Im SI, Shin SY, Na JO, Kim YH, Choi CU, Kim SH, Kim JW, Kim EJ, Han SW, Rha SW, Park CG, Seo HS, Oh DJ, Hwang C, Lim HE. Usefulness of neutrophil/lymphocyte ratio in predicting early recurrence after radiofrequency catheter ablation in patients with atrial fibrillation. Int J Cardiol. 2013 Oct 9;168(4):4398-400. doi: 10.1016/j.ijcard.2013.05.042. Epub 2013 May 28. No abstract available. PMID 23725815
- [Background] Ha AC, Wijeysundera HC, Birnie DH, Verma A. Real-world outcomes, complications, and cost of catheter-based ablation for atrial fibrillation: an update. Curr Opin Cardiol. 2017 Jan;32(1):47-52. doi: 10.1097/HCO.0000000000000348. PMID 27755137